CLINICAL TRIAL: NCT04369794
Title: COVID-19: BCG As Therapeutic Vaccine, Transmission Limitation, and Immunoglobulin Enhancement
Acronym: BATTLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Paulínia Municipal Hospital (Unknown)
Responsible Party: Principal Investigator, Leonardo Oliveira Reis, Professor Livre Docente, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-19 BATTLE trial
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Therapeutic Vaccine; BCG; SARS-CoV 2; Transmission
Keywords: BCG; Therapeutic Vaccine; COVID-19; SARS-CoV 2; Interferon Gamma; Immunoglobulin; Immunemodulation; Transmission
MeSH Terms: conditions — COVID-19 | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG vaccine (Active Comparator): BCG Group (n = 200): 0.1 ml of lyophilized, live, and attenuated BCG intradermal vaccine, containing between 2 and 8 x 1.000.000 C.F.U in a single dose.
  Interventions: Biological: BCG
- Placebo (Placebo Comparator): Placebo group (n = 200): 0.9% saline solution in the same volume as BCG vaccine in a single dose.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BCG — 0.1 ml of lyophilized, live and attenuated intradermal BCG vaccine, containing between 2 and 8 x 1.000.000 C.F.U in a single dose
  Other Names: Calmette Guerin bacillus
  Arms: BCG vaccine
Biological: Placebo — 0.9% saline in the same volume as the BCG vaccine in a single dose
  Arms: Placebo

SUMMARY:
To date, there is no vaccine or treatment with proven efficiency against COVID-19, and the transmissibility of the SARS-CoV-2 virus can be inferred by its identification in the oro-nasopharynx. The bacillus Calmette Guérin (BCG) has the potential for cross-protection against viral infections. This study evaluates the impact of previous (priming effect, from the titer of anti-BCG interferon-gamma) or current BCG exposure (boost with intradermal vaccine) on 1) clinical evolution of COVID-19; 2) elimination of SARS-CoV-2 at different times and disease phenotypes; and 3) seroconversion rate and titration (anti-SARS-CoV-2 IgA, IgM, and IgG).

DETAILED DESCRIPTION:
Prospective, randomized, double-blind, multicentre study with international design collaboration with central clinical and mechanistic outcomes with public health implications both epidemiological and therapeutic in the context of the pandemic of COVID-19, an emerging disease, which quickly disrupted health services including Brazil's Unified Health System (SUS), as well as the entire productive force and economy worldwide. Because it is recent, the basic evidence related to infection, such as incubation period, time of transmissibility, and seroconversion, is little known and the proposal's goals have the potential to redirect the vaccine. Exploring bacillus Calmette Guerin (BCG) that presents significant potential for immune activation, with recognized safety in decades of previous experience and clear potential in the context under analysis, with low cost and available, ensuring wide accessibility, especially in the context of SUS, on which it depends especially the most vulnerable portion of the Brazilian population, notably in the COVID-19 pandemic. Non-specific effects of BCG caused by monocyte epigenetic reprogramming may result in increased production of pro-inflammatory cytokines, conferring innate (trained) immunity and protection against viral infections, including SARS-CoV-2 with the potential to positively impact clinical evolution, viral elimination, and seroconversion of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age;
* laboratory or clinical-epidemiological confirmation of COVID-19 (history of close or home contact with a laboratory-confirmed case who has fever or at least one of the respiratory signs or symptoms, in the last 14 days after contact, and for which it was not possible to carry out the specific laboratory investigation)

Exclusion Criteria:

* Immunosuppressed patients of any kind;
* Pregnant women;
* More than 14 days from the onset of symptoms;
* Not accept participation or non-signature of the IC;
* Undiagnosed cases, suspected or probable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Clinical evolution of COVID-19 | 45 days of symptoms onset or diagnosis
  Classified as mild, moderate and severe
SARS-CoV-2 elimination | 7 days of symptoms onset or diagnosis
  Virus detection by PCR
Seroconversion rate and titration | 7 days of symptoms onset or diagnosis
  Titration of anti SARS-CoV-2 IgA, IgM and IgG

SECONDARY OUTCOMES:
Local and systemic adverse events to BCG vaccination | 3 months
  Classified according to type and severity

OTHER OUTCOMES:
SARS-CoV-2 elimination | 21 days of symptoms onset or diagnosis
  Virus detection by PCR
Seroconversion rate | 21 days of symptoms onset or diagnosis
  Titration of anti SARS-CoV-2 IgA, IgM and IgG
SARS-CoV-2 elimination | 45 days of symptoms onset or diagnosis
  Virus detection by PCR
Seroconversion rate and titration | 45 days of symptoms onset or diagnosis
  Titration of anti SARS-CoV-2 IgA, IgM and IgG

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo O Reis, MD, PhD, Principal Investigator — UroScience, University of Campinas
Locations (1):
- Hospital das Clínicas Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jalalizadeh M, Leme PAF, Buosi K, Dionato FAV, Dal Col LSB, Giacomelli CF, Reis LO. Healthcare Workers (HCWs) and non-HCWs reaction to Bacillus Calmette-Guerin (BCG) in the BATTLE trial. Vaccine. 2023 Oct 20;41(44):6599-6606. doi: 10.1016/j.vaccine.2023.09.031. Epub 2023 Sep 22. PMID 37743116
- [Derived] Dionato FAV, Jalalizadeh M, Buosi K, Visacri MB, Dal Col LSB, Giacomelli CF, Leme PAF, Maia CL, Moriel P, Reis LO. BCG vaccine safety in COVID-19 convalescent adults: BATTLE a randomized controlled trial. Vaccine. 2022 Jul 30;40(32):4603-4608. doi: 10.1016/j.vaccine.2022.06.039. Epub 2022 Jun 20. PMID 35738969
- [Derived] Jalalizadeh M, Buosi K, Dionato FAV, Dal Col LSB, Giacomelli CF, Ferrari KL, Pagliarone AC, Leme PAF, Maia CL, Yadollahvandmiandoab R, Trinh QD, Franchini KG, Bajgelman MC, Reis LO. Randomized clinical trial of BCG vaccine in patients with convalescent COVID-19: Clinical evolution, adverse events, and humoral immune response. J Intern Med. 2022 Oct;292(4):654-666. doi: 10.1111/joim.13523. Epub 2022 Jun 3. PMID 35599154